CLINICAL TRIAL: NCT07273032
Title: Clinical Application Research of Combined Therapy in ERAS for Accelerated Orthopedic Rehabilitation
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY2025PJ202
Record Dates: First submitted 2025-07-31; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-07

CONDITIONS: Meniscus Injury
Keywords: Patients who have undergone meniscus repair surgery under knee arthroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blank control group (Sham Comparator): Underwent meniscus plasty under knee arthroscopy
  Interventions: Procedure: Blank control group
- Lower limb rehabilitation training system combined with Henggu bone Injury Healing Agent interventio (Experimental): On the basis of undergoing meniscus formation surgery under knee arthroscopy, systematic intervention of lower limb rehabilitation training was received. After discharge, remote guidance for home rehabilitation was provided, and at the same time, Henggu bone Injury Healing Agent was started to be taken.
  Interventions: Procedure: Blank control group; Drug: Henggu Bone Injury Healing Agent Intervention Group; Device: Lower limb rehabilitation training system intervention group
- Henggu Bone Injury Healing Agent Intervention Group (Experimental): Patients received Henggu Bone Healing Formula concurrently after undergoing arthroscopic meniscal plasty.
  Interventions: Procedure: Blank control group; Drug: Henggu Bone Injury Healing Agent Intervention Group
- Lower limb rehabilitation training system intervention group (Experimental): On the basis of undergoing meniscus formation surgery under knee arthroscopy, systematic intervention of lower limb rehabilitation training was received, and remote guidance for home rehabilitation was provided upon discharge.
  Interventions: Procedure: Blank control group; Device: Lower limb rehabilitation training system intervention group

INTERVENTIONS:
Procedure: Blank control group — Underwent meniscus plasty under knee arthroscopy
Drug: Henggu Bone Injury Healing Agent Intervention Group — Patients received Henggu Bone Healing Formula concurrently after undergoing arthroscopic meniscal plasty.
  Arms: Henggu Bone Injury Healing Agent Intervention Group; Lower limb rehabilitation training system combined with Henggu bone Injury Healing Agent interventio
Device: Lower limb rehabilitation training system intervention group — On the basis of undergoing meniscus formation surgery under knee arthroscopy, systematic intervention of lower limb rehabilitation training was received, and remote guidance for home rehabilitation was provided upon discharge.
  Arms: Lower limb rehabilitation training system combined with Henggu bone Injury Healing Agent interventio; Lower limb rehabilitation training system intervention group

SUMMARY:
The double-blind method is adopted.Case selection Patients who underwent meniscus repair surgery under knee arthroscopy at Li Huili Hospital Affiliated to Ningbo University, the 906th Hospital of the People's Liberation Army (Joint Logistic Support Force of the Chinese People's Liberation Army), and Yangming Hospital Affiliated to Ningbo University (Yuyao People's Hospital), with ages set at 20 to 65 years old, are planned to be included in a sample size of 120 cases based on previous research experience, divided into 4 groups. They were respectively: the blank control group, the Henggu Bone Injury Healing Agent intervention group, the lower limb rehabilitation training system intervention group, and the Henggu Bone injury Healing agent combined with the lower limb rehabilitation training system intervention group, with 30 cases in each group. Grouping was conducted using a double-blind method, with random grouping carried out by a third-party organization.

1. Inclusion criteria: (1) The patient is conscious and aware of the content of this study; (2) Those with good compliance; (3) Possess good language communication skills.
2. Exclusion criteria: (1) Severely obese patients; (2) People with cognitive dysfunction; (3) Those with relevant serious complications; (4) Those with severe heart, liver or kidney insufficiency.
3. Exclusion criteria: Those who received intervention with other anti-inflammatory and analgesic drugs after the operation.

Criteria for terminating the study: Postoperative complications such as joint infection and deep vein thrombosis of the lower extremities occur after the operation.

Blank control group: No intervention measures Lower limb rehabilitation training system intervention group: Received rehabilitation system intervention after the operation Henggu Bone Injury Healing Agent Intervention Group: Take Henggu Bone Injury Healing Agent after the operation The combined intervention group: After the operation, they took Henggu bone injury Healing Agent and received rehabilitation system intervention The knee joint function and pain scores of each group, the implementation of the recovery plan, remote guidance of the rehabilitation system (applicable to the intervention group), and the duration of drug use: a total of 6 weeks of Henggu Bone Injury Healing Agent were evaluated at 1 day, 4 weeks, 3 months, and 6 months after the operation.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients with meniscus injury were conscious and aware of the content of this study. (2) Good compliance and cooperation with relevant drug treatments; (3) Possess good language communication skills.

Exclusion Criteria:

Patients with severe obesity; (2) People with cognitive dysfunction (such as Alzheimer's disease); (3) Those with severe heart, liver or kidney insufficiency.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS score, Limb symmetry index (LSI), HSS score, Lysholm score, International Knee Documentation Committee Knee Score (IKDC score), range of motion (ROM). | The first day after the operation, 4 weeks after the operation, 3 months after the operation, and 6 months after the operation.
  1.Visual Analogue Scale (VAS)Range: 0-10 points,Interpretation: 0 = no pain, 10 = worst possible pain.Directionality: Higher scores indicate more severe pain (worse outcome).2.Limb Symmetry Index (LSI)Range: 0-100%.Directionality: Higher scores indicate better limb symmetry (better outcome).3.Hospital for Special Surgery Knee Score (HSS)Range: 0-100 points,Directionality: Higher scores indicate better function (better outcome).4.Lysholm Knee Scoring ScaleRange: 0-100 points.Directionality: Higher scores indicate better knee function (better outcome).5.International Knee Documentation Committee Knee Score (IKDC)Range: 0-100 point,Directionality: Higher scores indicate better knee function (better outcome).6.Range of Motion (ROM)Range:0°-135°,Directionality: Higher values indicate greater mobility (better outcome).

IPD SHARING:
Plan to Share IPD: No